CLINICAL TRIAL: NCT03924817
Title: Registry Study on Prescription, Patient Pathways, Therapy Efficacy and Usage of Mandibular Advancement Devices in Obstructive Sleep Apnea - PATT-OSA Registry
Acronym: PATT-OSA
Status: Recruiting | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: PATT-OSA_Reg_07082023
Record Dates: First submitted 2019-03-26; First posted 2019-04-23 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During sleep, the muscle tonus in the oropharyngeal space is lost, the tongue might fall back andthe volume of the pharynx decreases. Air cannot pass through as it would in the awake state and thus airflow limitations occur. The person asleep might compensate the flow limitation by breathing faster, which causes the soft tissue to vibrate (= snoring). Further narrowing of the airways can lead to obstructive apneas (complete airway collapse and stopping of airflow). First line therapy for obstructive sleep apnea (OSA) is positive airway pressure (PAP) that keeps the airways open with a pneumatic splint. Since PAP involves wearing a facial mask that applies air pressure into the airways, some patients cannot tolerate this therapy. These patients might be candidates for an alternative treatment approach with a mandibular advancement device (MAD).

DETAILED DESCRIPTION:
During sleep, the muscles in the oropharyngeal space relax, the tongue falls back and the volume of the pharynx decreases. Air cannot pass through as it would in the awake state and thus airflow limitations occur. Diminishing airflow can lead to snoring or to the airways collapsing completely (obstructive sleep apnea, OSA). Patients who suffer from OSA have trouble breathing during sleep and will have a disturbed sleep architecture as repeated airway closure causes wake reactions and arousals. This does not only lead to severe daytime sleepiness with high risk of causing car accidents, for instance, but also affects synaptic activity during sleep and the balance of blood gas levels. These factors can have a aggravating effect on blood pressure and worsen the prognosis for cardiovascular comorbidities. First line therapy for obstructive sleep apnea (OSA) is positive airway pressure (PAP) that keeps the airways open with a pneumatic splint. Positive airway pressure is being applied through a facial mask and some patients cannot tolerate this therapy or refuse it. An alternative treatment approach is by fitting an MAD that the patient wears during sleep. An MAD pushes the lower jar forward and thereby increases the volume of the upper airways, thus preventing them to close. Studies have shown good compliance with MAD therapy and benefits in terms of sleepiness and quality of life. The Narval registry study aims to investigate MAD usage in real life and reasons for non-compliance. The registry aims to record patient characteristics (e.g. comorbidities) and side effects that lead to a termination of therapy, but also how the costs for therapy are split between the patient and public or private health insurance providers and how this affects therapy initiation and usage.

ELIGIBILITY:
Inclusion Criteria:

* Prescription of any mandibular advancement device
* Age ≥ 18 years
* Ability to understand the study information and information on usage of personal data
* Signed and dated informed consent

Exclusion Criteria:

* Patients with central sleep apnea (central AI > 5/hour)
* Patients with loose teeth and severe parodontitis
* Patients with completely missing teeth or removable tooth replacement, or with a teeth health insufficient to retain an MAD Patients with missing molars Patients with maximum protrusion of less than 5mm

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible for recruitment are male and female patients of ≥ 18 years who have been diagnosed with OSA and who are not eligible for PAP treatment (no tolerance of PAP therapy, therapy refusal for any reason). Patients who have been prescribed an MAD as treatment for OSA. Patients will be followed in their clinical routine treatment pathway.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of the Apnoea-Hypopnea-Index (AHI) at baseline compared to a follow-up after 3 months | 3 months
  Changes in the number of apnoeas (cessation of airflow) and hypopneas (reduced airflow) at baseline and at follow-up

SECONDARY OUTCOMES:
Changes in sleep-related quality of life from baseline compared to 3 months follow-up | 3 months
  Changes in sleep-related quality of life assessed with the questionnaire FOSQ (Functional Outcomes of Sleep Questionnaire). The Functional Outcomes of Sleep questionnaire is a "self-report measure designed to assess the impact of disorders of excessive sleepiness on multiple activities of daily living" (Weaver 1997). It consists of 10 questions categorized as General Productivity, Social Outcome, Activity Level, Vigilance, Sexual Activity. The range of scores for any item is 1-4. The potential range of scores for the total score is 5-20, with 5 meaning bad sleep-related quality of life and 20 good sleep-related quality of life. The total score is being calculated by calculating the mean of the subscale scores and then multiply that mean by five. Missing or not applicable answers will not be added when calculating the mean subscale scores.
Changes in daytime sleepiness from baseline compared to 3 months follow-up | 3 months
  Changes in daytime sleepiness assessed with the Epworth Sleepiness Scale questionnaire (ESS, measures the likelihood of a patient of falling asleep during daytime as self-reported outcome). The ESS is self-reported measure to assess whether a person would be prone to fall asleep in typical daily situations. It consists of 8 questions that can be answered with 0 = would never fall asleep, 1 = slight probability of falling asleep, 2 = moderate probability of falling asleep, 3 = high probability of falling asleep. The scores will be added up to give a total ranging from 0 - 24 and indicating different levels of excessive daytime sleepiness (6-10 higher than normal; 11-12 mild; 13-15 moderate; 16-24 severe).
Changes in snoring from baseline compared to 3 months follow-up | 3 months
  Changes in snoring assessed with a snoring questionnaire (the Thornton Snoring Scale contains 5 questions about snoring as subjective patient's measure). The Thornton Snoring Scale consists of 5 questions that can be answered with 0 = never, 1 = infrequently, 2 = frequently, 3 = most of the time. The scores will be added and when the sum of all answers is higher than 5, a snoring problem is indicated.
Usage of the MAD (mandibular advancement device) | 3 months
  Patients will be asked about how long and on how many days they were using the Narval MAD during the follow-up period. Patients will be offered a choice between "usage in total" - every night, 3-4 times a week, 1-2 times a week. Usage per night: Less than 1 hour, 1-3 hours, 4-5 hours.
Side effects with use of the MAD (mandibular advancement device) | 3 months
  Patients will be asked if they experienced side effects and which kind of side effects: Temporomandibular joint pain, dental pain, hypersalivation, dry mouth, local irritation, inflammation, dental fracture, broken MAD/device defect.
Document comorbidities of enrolled patients | 3 months
  Patients will be asked for relevant comorbidities (diabetes, hypertension, heart failure)
Remuneration of a MAD | 3 months
  Patients will be asked whether they bought the MAD themselves or if a public or private healthcare insurance provider paid the expenses
Satisfaction with therapy | 3 months
  Patients will be asked to rate their satisfaction with therapy on a scale of 1 (bad) to 10 (very good).
Document sleep disorders of enrolled patients | 3 months
  Sleep disorders will be recorded with a polygraphy or polysomnography (obstructive sleep apnoea, central sleep apnoea)
Continuation of therapy | 3 months
  Patients will be asked if they are going to continue therapy. Reasons for therapy termination shall be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schoebel, Prof, Principal Investigator — Ruhrlandklinik Essen
Locations (4):
- Germany (4):
  - Schlaf- und Beatmungszentrum Blaubeuren, Blaubeuren Abbey, Badden-Württemberg
  - Ruhrlandklinik Essen, Essen, North Rhine-Westphalia
  - Zentrum für Schlafmedizin Dr. Warmuth, Berlin
  - Universitätsklinikum Regensburg - Klinik für Innere Medizin II, Regensburg